CLINICAL TRIAL: NCT05226546
Title: Effectiveness and Safety of Platelet Rich Plasma (PRP) on Persistent Olfactory Dysfunction Related to COVID-19: Towards a New Therapeutic Hope
Brief Title: Effectiveness and Safety of Platelet Rich Plasma (PRP) on Persistent Olfactory Dysfunction Related to COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0762021210228
Record Dates: First submitted 2022-02-03; First posted 2022-02-07 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Anosmia; COVID-19
Keywords: PRP; Anosmia; COVID-19
MeSH Terms: conditions — Anosmia; COVID-19 | interventions — Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Patient underwent simple olfactive training for one month.
  Interventions: Other: olfactory training
- PRP injected group (Experimental): Patient had one injection in each olfactory cleft.
  Interventions: Drug: Platelet rich plasma (PRP)

INTERVENTIONS:
Drug: Platelet rich plasma (PRP) — PRP injections were performed in each olfactory cleft by nasal endoscopy and under local anesthesia, a sniffing stick test was performed before the injection and one month after
  Arms: PRP injected group
Other: olfactory training — The investigators compare the result of the PRP group to a control group how underwent simple olfactive training for one month.
  The control group matched for age, gender and olfactory score at baseline. The patients had a sniffing stick test at the beginning and also after one month of olfactory training.
  Arms: control group

SUMMARY:
Olfactory dysfunction (OD) is a well know symptom of coronavirus disease 2019 (COVID-19), accounting for 48 to 85% of patients. In 1 to 10% of cases, patients develop a chronic olfactory dysfunction (COD,) lasting more than 6 months. Recently, platelet-rich plasma (PRP) was used in patients with non-COVID-19 COD and authors reported encouraging results. In the present study, the investigators investigated the usefulness and safety of PRP injection in 56 patients with COVID-19 COD.

Our results showed that PRP in the olfactory cleft can increase the olfactory threshold one month after the injection. Moreover, our results suggest that timing of treatment may be an important factor and that PRP is a safe treatment because no adverse effects were reported throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Patient chronic olfactory dysfunction lasting more than 6 months after an infection of COVID-19

Exclusion Criteria:

* Patient under 18 years old
* Patient with blood disorder
* Blood thinner user
* Patient with abnormal findings on nasal endoscopy (e.g., polyposis, rhinosinusitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
efficity of 1 injection of PRP by Sniffing Sick test compare to a simple olfactory training | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Horoi, PhD, Study Director — CHU saint Pierre de Bruxelle
Locations (1):
- CHU saint pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steffens Y, Le Bon SD, Lechien J, Prunier L, Rodriguez A, Saussez S, Horoi M. Effectiveness and safety of PRP on persistent olfactory dysfunction related to COVID-19. Eur Arch Otorhinolaryngol. 2022 Dec;279(12):5951-5953. doi: 10.1007/s00405-022-07560-y. Epub 2022 Jul 29. PMID 35904632